CLINICAL TRIAL: NCT00465764
Title: Pilot Tolerance and Bone Status of Healthy, Term Infants Fed Infant Formulas
Brief Title: Tolerance and Development of Healthy, Term Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK44
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: healthy infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protein formula (Experimental): Feed as per HCP direction
  Interventions: Other: Alternate protein infant formula
- Standard infant formula (Active Comparator): Feed as per HCP instructions
  Interventions: Other: Standard infant formula

INTERVENTIONS:
Other: Alternate protein infant formula — Feed as per HCP directions
  Arms: Protein formula
Other: Standard infant formula — Feed as per HCP directions
  Arms: Standard infant formula

SUMMARY:
To compare the tolerance and early bone status of healthy, term infants fed formulas during the first three months of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants;
* Age 0-8 days of age;
* Exclusively formula fed;
* No use of vitamin/mineral supplements.

Exclusion Criteria:

* Maternal, fetal or perinatal medical history thought to have potential for negative effects on tolerance, growth or development.

Ages: 1 Day to 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean rank stool consistency at 14 days of age | 14 days of age

SECONDARY OUTCOMES:
Blood chemistries, bone mineral content, percent of feedings with spit-up or vomit associated with feeding | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Marlene W Borschel, PhD, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Children's Nutrition Research Center, Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831